CLINICAL TRIAL: NCT04918966
Title: Automatic Clinical Information Extraction Technology Development and Database Construction for Cardio-Vascular Emergency Patients Based on Voice and Image Recognition Technology
Brief Title: Development of Cardio-Vascular Emergency Patients Database Using Voice and Image Technology
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Collaborators: National Research Foundation of Korea (Other)
Responsible Party: Sponsor
Other Study IDs: SNUEMSAVCV
Record Dates: First submitted 2021-06-01; First posted 2021-06-09 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-05

CONDITIONS: Cardiovascular Diseases
Keywords: Image recognition; Voice recognition; Emergency department
MeSH Terms: conditions — Cardiovascular Diseases; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Video and audio data of cardio-vascular patients who visit the emergency department (ED) will be collected to build a database. Clinical information retrieved from the database using voice and image technology will be compared to that retrieved by physicians. The degree of agreement will be evaluated.

DETAILED DESCRIPTION:
Study Objectives:

1. To develop a platform to record video and audio data of cardio-vascular patients who visited the ED.
2. To retrieve clinical information using voice and image technology.
3. To develop a tool to retrieve clinical information using voice and image technology.
4. To build a clinical database using video and audio data using voice and image technology.

Study design: Single-center observational study (tertiary hospital emergency department in Korea).

A platform to record video and audio data of physicians examining patients will be developed. The camera and microphone will be installed at an optimal location to retrieve video and audio data of cardio-vascular patients.

Voice and image technology will be used to retrieve clinical information including chief complaint, type and onset of symptoms, past medical history, and physical examination results to build a database. Clinical information including examination notes, diagnosis, patient vital signs, test results, and ED results will be retrieved from the hospital database.

ELIGIBILITY:
Inclusion Criteria:

* Age 19 years or older
* Visited the emergency department of the study hospital
* Chief complaint of chest pain, dyspnea, syncope, altered mentality, side weakness, dizziness, and dysarthria

Exclusion Criteria:

* Patients who do not agree to enroll to this study
* Pregnant patient
* Without a family
* Foreign patients

Min Age: 19 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adults who visit the emergency department with cardio-vascular chief complaints and without one of the exclusion criteria will be enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2018-08-07 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
The degree of agreement between clinical information retrieved using voice/image technology and information recorded by physicians. | At the time of study completion (March 2023 anticipated).
  Clinical information include chief complaint, type and onset of symptoms, and physical examination results.

CONTACTS AND LOCATIONS:
Overall Officials: Ki Jeong Hong, PhD, Study Director — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea